CLINICAL TRIAL: NCT04673968
Title: Efficacy of Prehabilitation on Fitness, Surgical Outcomes and Mitochondria Functionality in Patients With Esophageal Cancer Undergoing Neoadjuvant Chemotherapy
Brief Title: Prehabilitation on Fitness, Surgical Outcomes and Mitochondria Functionality in Patients With Esophageal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 201901758B0
Record Dates: First submitted 2020-11-24; First posted 2020-12-17 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2022-08

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Preoperative Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- prehabilitation (P) (Active Comparator): inhospital exercise training 5 times/week, 5~6 weeks during nCRT (neoadjuvant chemoraiotherapy); home exercise 5 times/week, 5~6 weeks, between completion of nCRT and before surgery
  Interventions: Other: prehabilitation
- control group (C) (No Intervention): no prehabilitation

INTERVENTIONS:
Other: prehabilitation — inhospital exercise training 5 times/week, 5~6 weeks during nCRT; home exercise 5 times/week, 5~6 weeks, between completion of nCRT and before surgery
  Arms: prehabilitation (P)

SUMMARY:
The most often reported complications of patients with resectable esophageal malignancies are pulmonary (25~57%), which may cause increased intensive care unit utilization, prolonged length of hospital stay, increased mortality and medical expense. Also, neoadjuvant chemotherapy has a deleterious effect on patients' cardiopulmonary capacity, strength and muscle mass. Prehabilitation includes preoperative exercise training and nutrition management. The reporting outcome regarding whether it improves surgical outcomes is inconsistent. One of the reasons is that pulmonary complication tends to occur in patients with low cardiopulmonary fitness, but all studies included patients with all level of fitness.

Most of the chemotherapy interferes with cell division to inhibit tumor growth but is also harmful to mitochondria functionality. For example, Cisplatin and Paclitaxel, commonly used in esophageal cancer, alter mitochondria function, caused by disruption of respiratory chain function and increased production of reactive oxygen species. However, it remains unclear their negative effects on the oxidative phosphorylation capacity of mitochondria (OXPHOS). Furthermore, whether prehabilitation reverses this negative effect is scarcely explored.

Patients will be inquired to participate and randomized into prehabilitation or control group. The latter will undergo conventional therapy only, while the former will receive additional prehabilitation program. The prehabilitation program encompasses supervised and home-based aerobic, resistance training (large and inspiratory muscle) and nutrition management. The supervised exercise training will be performed right before or after the radiotherapy. Outcome variables are fitness-related testing [the 1st year], quality of life and surgical outcomes [the 2nd year] and mitochondria functionality (OXPHOS, membrane potential, matrix oxidant burden) [the 3rd year]. Evaluation is performed 3 times at baseline, before surgery and 4 weeks after surgery.

DETAILED DESCRIPTION:
Neoadjuvant chemotherapy has significantly improved patient outcomes. The majority of patients with resectable esophageal malignancies are considered for neoadjuvant treatment. However, esophagectomy and chemotherapy have disadvantages. Morbidity and mortality associated with esophagus resection remain high. The most often reported complications are pulmonary (25~57%), which may cause increased intensive care unit utilization, prolonged length of hospital stay, increased mortality and medical expense.

Also, neoadjuvant chemotherapy has a deleterious effect on patients' cardiopulmonary capacity, strength and muscle mass. Prehabilitation includes preoperative exercise training and nutrition management. The reporting outcome regarding whether it improves surgical outcomes is inconsistent. One of the reasons is that pulmonary complication tends to occur in patients with low cardiopulmonary fitness, but all studies included patients with all level of fitness. In the current investigation, only those with low cardiopulmonary fitness will be enrolled.

Most of the chemotherapy interferes with cell division to inhibit tumor growth but is also harmful to mitochondria functionality. For example, Cisplatin and Paclitaxel, commonly used in esophageal cancer, alter mitochondria function, caused by disruption of respiratory chain function and increased production of reactive oxygen species. However, it remains unclear their negative effects on the oxidative phosphorylation capacity of mitochondria (OXPHOS). Furthermore, whether prehabilitation reverses this negative effect is scarcely explored.

This is a three-year prospective randomized trial. Patients who suffer from locally-advanced esophageal cancer and will receive neoadjuvant chemoradiotherapy and operation in Chang Gung Memorial Hospital at Linkou will be inquired to participate. A total of 160 patients will be recruited expectedly and randomized into prehabilitation or control group. The latter will undergo conventional therapy only, while the former will receive additional prehabilitation program. The prehabilitation program encompasses supervised and home-based aerobic, resistance training (large and inspiratory muscle) and nutrition management. The supervised exercise training will be performed right before or after the radiotherapy. Outcome variables are fitness-related testing (cardiopulmonary exercise testing, 6-minute walk distance, handgrip, and body composition, maximal inspiratory pressure and muscle oxidative capacity) [the 1st year], quality of life and surgical outcomes (length of stay in the hospital and intensive care unit, surgical complication, perioperative pulmonary complications and medical expense) [the 2nd year] and mitochondria functionality (OXPHOS, membrane potential, matrix oxidant burden) [the 3rd year]. Evaluation is performed 3 times at baseline, before surgery and 4 weeks after surgery.

The investigators hypothesize that prehabilitation increases functional reserve to improve surgical outcomes [2nd year] in a subpopulation of patients with esophageal cancer who receive neoadjuvant chemo-radiotherapy plus having low cardiopulmonary fitness. It also reverses fitness decline during neoadjuvant chemotherapy [1st year], partly through amelioration of mitochondria functionality [3rd year]. The goal of the investigation is to provide an applicable prehabilitation model and establish its efficacy at clinical, tissue and cellular levels.

ELIGIBILITY:
Inclusion Criteria:

* nonmetastatic esophageal cancer patients.
* V'O2 < 21ml/min/kg
* abnormality on spirometry.

Exclusion Criteria:

* Resting heart rate greater than 100 beats per minute
* Atrial fibrillation or flutter
* Poor control of high blood pressure or diabetes
* Patients with peripheral arterial occlusive disease
* Patients with end-stage renal disease
* Patients receiving anticoagulant therapy
* Neurological instability

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2020-02-25 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Exercise capacity of all participants by Cardiopulmonary Exercise Test (CPET) | three years
  Cardiopulmonary Exercise Test
Exercise capacity of fitness-related parameters: 6-minute walk distance | three years
  Detection of 6-minute walk distance in meters
Exercise capacity of fitness-related parameters: hand grip | three years
  Detection of hand grip strength in kilograms
Body composition | three years
  Body composition analysis

SECONDARY OUTCOMES:
Surgical outcomes of inpatient days | three years
  length of stay in the hospital and intensive care unit in days
Complications outcomes | three years
  Preoperative and surgical complications analysis
Mitochondria functionality | three years
  Mitochondrial function of lymphocytes

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Chun Huang, MD, PhD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan